CLINICAL TRIAL: NCT04695899
Title: Observational Study Evaluating Zirconia Dental Implants and Screw Retained Implant Crowns for Metal-free Single Tooth Replacement
Brief Title: Zirconia Implants for Replacement of a Single Tooth
Status: Active, not recruiting | Type: Observational
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-01434
Record Dates: First submitted 2021-01-04; First posted 2021-01-05 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Partial-edentulism
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Crevicular/sulcus fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Dental Implant — See Section "Procedures".

SUMMARY:
First, the surgical insertion of a ceramic (zirconia) dental implant will be performed in a single-tooth gap according to current state-of-the-art protocols. After a 3-months healing phase, a ceramic tooth replacement (a.k.a. implant crown) will be screw-retained on the implant and will be ready for full chewing, aesthetic and speech function.

DETAILED DESCRIPTION:
Surgery Implant placement will be performed according to a standardized, well-documented surgical protocol considered internationally as state-of-the art therapy for titanium implants since decades (Buser & von Arx 2000, Buser et al. 2004). In summary, an osteotomy will be performed in the edentulous bone under local anaesthesia and after the elevation of a full-thickness mucoperiosteal flap. The screw-shaped implant will then be inserted into the osteotomy. Particular emphasis will be set on risk minimization for adjacent anatomical structures (e.g. nerves, adjacent teeth), on sufficient primary implant stability, on circular embedding in > 1 mm thick bone walls and on correct three-dimensional implant positioning. In cases with insufficient bone volume, guided bone regeneration (GBR) will be performed using autogenous bone chips from the adjacent area, well-documented bovine bone mineral and resorbable porcine collagen membranes. The flaps will then be sutured around the implant healing cap (non-submerged healing). Primary flap closure will be preferred in cases with GBR (submerged healing). 12 ± 2 weeks after placement, submerged implants will be uncovered under local anaesthesia, then the osseointegration of the implants will be verified clinically and radiographically, and impressions will be taken.

Restoration Restoration in group A (tooth replacement in FDI positions 14 - 24): fixed implant-supported provisional for 3 months, then final restoration with all-ceramic screw-retained single implant-supported crown (abutment made of zirconium dioxide and crown finalized with hand-build up ceramic veneering material) Restoration in group B (tooth replacement in all other positions): all-ceramic screw-retained single implant-supported crown (abutment made of zirconium dioxide and monolithic lithium disilicate ceramic crown.

ELIGIBILITY:
Inclusion criteria (site level):

* partial edentulism (any FDI position between 17 and 47)
* healed extraction site (type 2, 3 or 4 implant placement) or native bone
* opposing dentition: natural teeth, fixed or removable restoration

Exclusion criteria (site level):

* inadequate ridge or gap dimensions for the test device (simultaneous bone augmentation allowed)
* lack of primary stability of the implant

Inclusion criteria (patient level):

* self-referred or on purpose referred patient requiring a metal-free, all-ceramic implant therapy
* age ≥18 years and ≤ 80
* capable of providing written informed consent and compliance to the protocol
* physical status PS1 and PS2 (American Society of Anesthesiologists).

Exclusion criteria (patient level):

* pregnancy or lactation
* inadequate oral hygiene
* untreated periodontitis or gingivitis
* mucosal diseases such as erosive lichen planus
* smoking habit with >5 cig/d
* severe bruxism or clenching habits
* uncontrolled diabetes or conditions resulting in or requiring immunosuppression, radiation, chemotherapy, frequent use of antibiotics or antiresorptive medication such as bisphosphonates

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: General population.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Survival Rate | 12 months
  How many implants are still in function

SECONDARY OUTCOMES:
Success Rate | 10 years
  How many implants satisfy current biological and technical success criteria

CONTACTS AND LOCATIONS:
Overall Officials: SImone FM Janner, PD Dr., Principal Investigator — University of Bern
Locations (1):
- University of Bern - Klinik für rekonstruktive Zahnmedizin und Gerodontologie, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No